CLINICAL TRIAL: NCT04895748
Title: A Phase I/Ib, Open-label, Multi-center Study of DFF332 as a Single Agent and in Combination With Everolimus or IO Agents in Patients With Advanced/Relapsed ccRCC and Other Malignancies With HIF2α Stabilizing Mutations
Brief Title: DFF332 as a Single Agent and in Combination With Everolimus & Immuno-Oncology Agents in Advanced/Relapsed Renal Cancer & Other Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDFF332A12101; 2024-513379-41 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Renal Cell
Keywords: ccRCC; RCC; Kidney; DFF332; NIR178; PDR001; RAD001; Everolimus; Spartalizumab; Taminadenant; Von Hippel-Lindau Disease; Hereditary leiomyomatosis and renal cell cancer syndrome; Paraganglioma; Pheochromocytoma
MeSH Terms: conditions — Carcinoma, Renal Cell; von Hippel-Lindau Disease; Hereditary leiomyomatosis and renal cell cancer; Paraganglioma; Pheochromocytoma | interventions — Everolimus; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1 Dose Escalation DFF332 (Experimental): DFF332 Single Agent
  Interventions: Drug: DFF332
- Arm 2 Dose Escalation DFF332 + Everolimus (Experimental): Combination treatment DFF332 + Everolimus. This arm will not open.
  Interventions: Drug: DFF332; Drug: RAD001
- Arm 3 Dose Escalation DFF332 + Spartalizumab + Taminadenant (Experimental): Combination treatment DFF332 + Spartalizumab + Taminadenant. This arm will not open.
  Interventions: Drug: DFF332; Drug: PDR001; Drug: NIR178
- Arm 1a Dose Expansion DFF332 in ccRCC (Experimental): DFF332 Single Agent in patients with ccRCC (age 18 years old and above). This arm will not open.
  Interventions: Drug: DFF332
- Arm 1b Dose Expansion DFF332 in HIF stabilizing malignancies (Experimental): DFF332 Single Agent in patients with HIF stabilizing malignancies (age 12 years old and above). This arm will not open.
  Interventions: Drug: DFF332
- Arm 2a Dose Expansion DFF332 + Everolimus in ccRCC (Experimental): Combination treatment DFF332 + Everolimus in patients with ccRCC (age 18 years old and above). This arm will not open.
  Interventions: Drug: DFF332; Drug: RAD001
- Arm 3a Dose Expansion DFF332 + Spartalizumab + Taminadenant in ccRCC (Experimental): Combination treatment DFF332 + Spartalizumab + Taminadenant in patients with ccRCC (age 18 years old and above). This arm will not open.
  Interventions: Drug: DFF332; Drug: PDR001; Drug: NIR178

INTERVENTIONS:
Drug: DFF332 — Hif2alpha inhibitor
Drug: RAD001 — mTOR inhibitor
  Other Names: Everolimus
  Arms: Arm 2 Dose Escalation DFF332 + Everolimus; Arm 2a Dose Expansion DFF332 + Everolimus in ccRCC
Drug: PDR001 — anti-PD-1
  Other Names: Spartalizumab
  Arms: Arm 3 Dose Escalation DFF332 + Spartalizumab + Taminadenant; Arm 3a Dose Expansion DFF332 + Spartalizumab + Taminadenant in ccRCC
Drug: NIR178 — Adenosine A2A antagonist receptor
  Other Names: Taminadenant
  Arms: Arm 3 Dose Escalation DFF332 + Spartalizumab + Taminadenant; Arm 3a Dose Expansion DFF332 + Spartalizumab + Taminadenant in ccRCC

SUMMARY:
This is first in human study of DFF332, a small molecule that targets a protein called HIF2α. By acting on HIF2α, DFF332 may be able to stop the growth of certain types of cancer. DFF332 will be tested at different doses as single agent and in combination with Everolimus (RAD001, an mTOR inhibitor), and also in combination with Spartalizumab (PDR001, an anti-PD1) plus Taminadenant (NIR178, an adenosine A2A receptor antagonist), in patients with advanced clear cell renal cell carcinoma and other malignancies with HIF stabilizing mutations.

DETAILED DESCRIPTION:
This is a first in human (FIH), Phase I/Ib, open-label, multi-center study of DFF332 as a single agent and in combination with Everolimus or Spartalizumab plus Taminadenant in patients with advanced clear cell renal cell carcinoma and other malignancies with HIF stabilizing mutations.

The study consists of two parts, dose escalation and dose expansion. The dose escalation part of the study will initially evaluate DFF332 single agent. Dose escalation groups receiving DFF332 in combination with Everolimus or DFF332 in combination with Spartalizumab plus Taminadenant will open after at least two dose levels of single agent DFF332 have been evaluated.

The dose expansion part of single agent will include two treatment arms: Arm1A will enroll ccRCC patients (age 18 yo or above) and Arm1B will enroll patients with malignancies harboring HIF stabilizing mutations (age 12 yo and above). These include the following:

* Malignancies with VHL mutations (e.g. Von Hippel-Lindau disease)
* Malignancies with FH mutations (e.g. Hereditary leiomyomatosis and renal cell carcinoma)
* Malignancies with mutations in SDHD, SDHAF2, SDHC, SDHB, SDHA (e.g. Hereditary paraganglioma and pheochromocytoma syndrome)
* Malignancies with EPAS1/HIF2A mutations
* Malignancies with ELOC/TCEB1 mutations

The expansion part of the combination therapies will enroll patients with ccRCC and include Arm2A (DFF332 with Everolimus) and Arm3A (DFF332 with Spartalizumab plus Taminadenant).

Novartis halted enrollment of study CDFF332A12101 in September 2023 due to business reasons and not due to safety concerns. The DFF332 single agent dose expansion arms and the dose escalation and expansion of the combination arms will not open.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years of age For Arm 1B: Male and female of age ≥ 12 years of age
2. Histologically confirmed and documented clear cell renal cell carcinoma (ccRCC). Disease must be measurable as determined by RECIST v1.1.

   For Arm 1B: histologically confirmed and documented malignancies in the context of the following cancer predisposing syndromes/disorders or harboring somatic mutations on one of these genes:
   * Malignancies with VHL mutations (e.g. Von Hippel-Lindau disease)
   * Malignancies with FH mutations (e.g. Hereditary leiomyomatosis and renal cell carcinoma)
   * Malignancies with mutations in SDHD, SDHAF2, SDHC, SDHB, SDHA (e.g. Hereditary paraganglioma and pheochromocytoma syndrome)
   * Malignancies with EPAS1/HIF2A mutations
   * Malignancies with ELOC/TCEB1 mutations Note: Mutations must have been previously identified through local molecular assays.
3. Patient with unresectable, locally advanced or metastatic ccRCC with documented disease progression following all standard of care therapy, including PD-1/L1 checkpoint inhibitor and a VEGF targeted therapy as monotherapy or in combination.

   Escalation: No restriction on the number of prior treatments Expansion (with the exception of Arm 1B): Up to 3 prior lines of treatment for advanced/metastatic disease For Arm 1B: Patients must have either metastatic disease or locally advanced disease that is unresectable or that patients be unfit for resection or other treatment modalities. Patients must have received prior standard therapy appropriate for their tumor type and stage of disease, and have no available therapies of proven clinical benefit; or in the opinion of the investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy.
4. For patients age ≥ 16 years: ECOG performance status ≤ 1 For patients age ≥ 12 and < 16 years: Lansky performance status ≥ 70

Exclusion Criteria:

1. History of seizure disorder & extrapyramidal (EPS) symptoms
2. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥ 2), uncontrolled hypertension
   * Patients with corrected QT using the Fridericia's correction (QTcF) > 470 msec for all patients on screening ECG or congenital long QT syndrome Acute myocardial infarction or unstable angina < 3 months prior to study entry
   * History of stroke or transient ischemic event requiring medical therapy
   * Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
3. Treatment with any of the following anti-cancer therapies prior to the first dose of study treatment within the stated timeframes:

   1. ≤ 4 weeks for radiation therapy or limited field radiation for palliation within ≤ 2 weeks prior to the first dose of study treatment.
   2. ≤ 4 weeks or ≤ 5 half-lives (whichever is shorter) for chemotherapy or biological therapy (including monoclonal antibodies) or continuous or intermittent small molecule therapeutics or any other investigational agent.
   3. ≤ 6 weeks for cytotoxic agents with major delayed toxicities, such as nitrosourea and mitomycin C.
   4. ≤ 4 weeks for immuno-oncologic therapy, such as CTLA-4, PD-1, or PD-L1 antagonists.
   5. Patients who have undergone major surgery ≤ 4 weeks prior to first dose of study treatment or who have not recovered for the surgical procedure.
4. Patient previously treated with a HIF2α inhibitor.
5. Uncontrolled concurrent illness including, but not limited to, ongoing active infection, uncontrolled hypertension, active peptic ulcer disease or gastritis, active bleeding diatheses, including any Patient known to have evidence of acute or chronic hepatitis B, hepatitis C, human immunodeficency virus (HIV), or a psychiatric illness/social situation that in the investigator's opinion would limit compliance with study requirements or compromise the ability of the patient to give written informed consent. Patients with chronic HBV or HCV disease that is controlled under antiviral therapy are allowed in the expansion parts but not in the escalation parts.
6. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
7. Presence of Grade ≥ 2 toxicity according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAEv5.0), from prior cancer therapy with the exception of neuropathy (inclusion of patients with neuropathy of Grade 2 or less is permitted), ototoxicity, and alopecia.
8. Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Number of participants with AEs/SAEs to characterize the safety and tolerability of DFF332 as a single agent, in combination with Everolimus (RAD001), and in combination with Spartalizumab (PDR001) plus Taminadenant (NIR178) in patients with advanced clear cell Renal Cell Carcinoma (ccRCC) and advanced malignancies with Hypoxia Inducible Factor (HIF) stabilizing mutations
Number of participants with dose interruptions and dose reductions | 3 years
  Number of participants with dose interruptions and dose reductions to characterize the tolerability of DFF332 as a single agent, in combination with Everolimus (RAD001), and in combination with Spartalizumab (PDR001) plus Taminadenant (NIR178) in patients with advanced ccRCC and advanced malignancies with HIF stabilizing mutations.
Dose intensity for DFF332 for dose escalation and expansion | 3 years
  Dose intensity will be computed as the ratio of actual cumulative dose received and actual duration of exposure
Incidence of Dose Limiting Toxicities (DLTs) in Cycle 1 (28 days) for DFF332 as a single agent and in combinations | 28 days
  Number of participants with DLTs

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 3 years
  To assess the anti-tumor activity of DFF332 as single agent and combination in patients with advanced ccRCC and with advanced malignancies with HIF stabilizing mutations based on RECIST v1.1
Best Overall Response (BOR) | 3 years
  To assess the anti-tumor activity of DFF332 as single agent and combination in patients with advanced ccRCC and with advanced malignancies with HIF stabilizing mutations based on RECIST v1.1
Progression Free Survival (PFS) for Recommended Dose (RD) only | 3 years
  To assess the anti-tumor activity of DFF332 as single agent and combination in patients with advanced ccRCC and with advanced malignancies with HIF stabilizing mutations based on RECIST v1.1
Duration of Response (DOR) for Recommended Dose (RD) Only | 3 years
  To assess the anti-tumor activity of DFF332 as single agent and combination in patients with advanced ccRCC and with advanced malignancies with HIF stabilizing mutations based on RECIST v1.1
Disease Control Rate (DCR) | 3 years
  To assess the anti-tumor activity of DFF332 as single agent and combination in patients with advanced ccRCC and with advanced malignancies with HIF stabilizing mutations based on RECIST v1.1
Maximum Concentration (Cmax) of DFF332 single agent and combination | 3 years
  PK parameters will be based on plasma concentration of DFF332 and Taminadenant, whole blood concentration of Everolimus, serum concentration of Spartalizumab
Area under the concentration-time curve (AUC) of DFF332 single agent and combination | 3 years
  PK parameters will be based on plasma concentration of DFF332 single agent and in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (5):
  - City of Hope National Medical, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - WA Uni School Of Med, St Louis, Missouri
  - Memorial Sloane Ketterin Cancer Ctr, New York, New York
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, Brno, Czechia
- Novartis Investigative Site, Villejuif, France
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No